CLINICAL TRIAL: NCT02428803
Title: Interactive Videoconferencing in the Provision of Remote Peritoneal Dialysis
Acronym: Telemedicine
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Eric Wallace, Assistant Professor Medicine - Nephrology, University of Alabama at Birmingham
Other Study IDs: X141112004
Record Dates: First submitted 2015-04-21; First posted 2015-04-29 (Estimated); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: ESRD
Keywords: Peritoneal Dialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Telemedicine

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Telemedicine — Patients will be administered the KDQOL-SF and the IIRS and will all start in the standard of care arm. During this time period the patients will receive 6 months of visits as per the usual standard of care. At the end of 6 months the KDQOL-SF and IIRS will again be administered. The patient will then transition to the telemedicine arm of the study for the duration of 6 months. During this time, the patient will come to the dialysis unit on a quarterly basis for a standard visit with labs being drawn in-center and for an in-center Kt/V. For the 2 months following the visit ,however, the patient will not be required to come to the dialysis unit. The monthly face to face and labs will be achieved remotely

SUMMARY:
Home dialysis patients must be seen in a face to face visit on a monthly basis. For patients who live remotely these visits may impact their quality of life due to the amount of time needed to attend these visits. The central hypothesis is that implementation of telemedicine visits as a substitute for the 2 out of 3 monthly face-to-face visits over a 6 month period will improve quality of life as judged by the quality of life (QoL) indices Kidney Disease Quality of Life - Short Form and the Illness Intrusiveness Ratings Scale when compared to QoL scales taken during a time period when the patient is on standard of care.

DETAILED DESCRIPTION:
Background:

Peritoneal Dialysis is used by over 100,000 patients worldwide but only about 7% of patients in the United States. 1 As it is much less expensive than its in-center hemodialysis counterpart and provides improved quality of life, strategies are needed to increase its utilization. One potential barrier to peritoneal dialysis is the geographic barriers to care which exist in geographically diverse and large countries such as Canada, India, Australia, and the United States. 2,3 Access to an experienced home dialysis unit is limited in many parts of the United States and can contribute to low utilization rates by physician discomfort with the therapy as well as increased technique failure rates with inexperienced centers. 4-7 Prakash et al recently have shown that only 55% of dialysis units are certified to provide home dialysis. 8 In more rural networks such as network 8 (Alabama, Mississippi, and Tennessee), this number drops to 38% thus increasing the geographic barriers to the provision of home dialysis care. Patients currently living in rural areas and on a home therapy are faced with long commutes and time commitments adding up to significant financial hardships for the patients. Furthermore, these commutes impact quality of life. Telemedicine and telemonitoring may provide a means to bridge these geographic barrier thus improving access to home dialysis care and improving patient quality of life on the therapy and thus increasing its utilization.

The use of telemedicine in the provision of home dialysis care has received very limited attention worldwide and even less in the United States. Early studies using telemedicine in remote care suffered from high costs of implementing secure T1 lines and limited technology.9 Gallar et al in Spain published 2 years of experience using alternating videoconferencing visits and standard hospitalized visits, showing cost savings, ability to evaluate the patient for edema and exit site evaluation, as well as decreased time associated with each visit. 10 Nakamoto et al. in Japan published on their tool to transmit blood pressures, glucose readings remotely etc. 11 Since these initial studies and conceptualization of telemedicine, technology has increased at a very fast pace. Videoconferencing technology has become much smaller, more sophisticated, easier to use, and more inexpensive making it a mainstay in daily life including applications such as face time and skype. Technology literacy as well has continued to increase since early 2000. A recent survey among peritoneal dialysis patients showed that 88% owned a computer and 94% knew how to use a computer. 12 Furthermore, 83% of patients wished to participate in telemedicine. 12 It is within this environment that telemedicine and the application to home dialysis may begin to transform the delivery of care in home dialysis thus increasing peritoneal dialysis utilization by improving convenience of the therapy and improving the quality of life. Such interventions are already gaining popularity in countries such as India. 3 Studies are needed to determine the feasibility of telemedicine in the provision of home dialysis care in the United States and if quality of life of patients using this mechanism are improved. Furthermore, studies showing outcomes are similar if not improved using telemedicine are needed.

The long-term goal of this project is to improve access to peritoneal dialysis care and the quality of lives of patients on dialysis by evaluating ways to eliminate the geographic barrier. The objective here is to determine if specifically telemedicine has this capacity. By evaluating and establishing a framework by which home dialysis care could be provided via telemedicine and determining the impact on quality of life for these patients, policy could be informed as to coverage of telemedicine as a substitute for the current face-to-face requirement by Medicare. Furthermore, this intervention has the possibility of improving quality of life and if effective possibly increasing the utilization of peritoneal dialysis both by patients rural and urban due to increased convenience of the therapy with respect to in-center hemodialysis. The central hypothesis is that implementation of telemedicine visits as a substitute for the 2 out of 3 monthly face-to-face visits over a 6 month period will improve quality of life as judged by the quality of life (QoL) indices Kidney Disease Quality of Life - Short Form and the Illness Intrusiveness Ratings Scale when compared to QoL scales taken during a time period when the patient is on standard of care.

Specific Aims

1. Determine the impact of telemedicine on quality of life as indicated two quality of life surveys: 1) The KDQOL- SF and the Illness Intrusiveness Ratings Scale .

   The investigators postulate that patients, during the telemedicine intervention will improve the quality of life scores on the KDQOL-SF form by the minimum clinically significant change of 3 points, as compared to themselves during a time period of standard of care visits (Not telemedicine).
2. Determine the feasibility of the use of telemedicine and remote monitoring in the provision of care for peritoneal dialysis patients as a substitute for two out of 3 monthly face-to-face visits over a 6 month period.

   Based on the work by Nayak et al. in India, the investigators feel that telemedicine visits as a substitute for the face-to-face visit will be both feasible and advantageous.
3. Obtain preliminary data on efficacy of the intervention with regards to outcomes with a composite endpoint of episodes of peritonitis and hospitalizations.

The investigators postulate that there will be either no difference in outcomes or an improvement in outcomes in the telemedicine intervention arm.

Study Design:

Patients will be recruited from the University of Alabama at Birmingham Peritoneal Dialysis Unit. All patient's addresses are known and will be screened in order to determine inclusion criteria. Upon enrollment, patients will be administered the KDQOL-SF and the IIRS. Patient will all start in the standard of care arm. During this time period the patients will receive 6 months of visits as per the usual standard of care. Data will be collected during this time regarding hospitalizations, peritonitis, technique failures, and access procedures. Monthly labwork including hemoglobin, phosphorus, parathyroid level, iron, total iron binding capacity, and ferritin will also be collected. At the end of 6 months the KDQOL-SF and IIRS will again be administered.

The patient will then transition to the telemedicine arm of the study for the duration of 6 months. During this time, the patient will come to the dialysis unit on a quarterly basis for a standard visit with labs being drawn in-center and for an in-center Kt/V. For the 2 months following the visit ,however, the patient will not be required to come to the dialysis unit. The monthly face to face and labs will be achieved remotely.

In order to do this, the investigators have partnered with the Alabama Department of Public Health. During the telemedicine visits, the patient will present to their county health department which are now outfitted with the capability to provide interactive telemedicine visits.

Exam: The patient will be examined during this telemedicine encounter using blue-tooth stethoscopes, placed on the patients chest by personnel in the county health department. The exit site will be examined using the remote camera. Fluid status will be monitored by both lung exam, weights which the patient does on a routine basis, and the examination of pitting edema as done over a telemedicine interface.

Labs- On the quarterly "standard" visit during the telemedicine intervention, the patient will be given 2 preaddressed and prestamped containers with all vials needed to collect their monthly labs. The patient during their telemedicine visits will bring this container with blood collection tubes to the county health department. There, personnel a the health department will perform phlebotomy, using the predetermined blood collection tubes. Once filled, these tubes will be sent in the prestamped container to the Davita Central Lab for further processing. In this way, no additional cost for labs will be incurred, and lab results will be standardized in one central lab.

Flow sheets: Patients records of therapy will be obtained using the Baxter ProCard. The patient will be trained on these cards prior to going to the telemedicine arm of the study. The patients will then be given 2 cards. Patients will use 1 procard for the month, and prior to their telemedicine visit will send this card in for download. Patients will then begin to use thesecond card, the previous card will be sent back to the patient via mail prior to their second visit such that it is had for their 3rd month.

Remote QoL Surveys: Patients will be administered either over the phone or on a paper form depending on literacy the KDQOL-SF and the IIRS survey on Visit 3, and Visit 6.

After completion of telemedicine arm, patients will return to Standard of Care and after 2 months of being back on standard of care, KDQOL-SF and IIRS again will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 or greater
* On Peritoneal Dialysis
* Living in a different county than that of the UAB Home Dialysis Unit ( Any county other than Jefferson County)
* Patients have to be stable on therapy for 2 months prior to enrollment

Exclusion Criteria:

* Living in Jefferson County

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: UAB patients on peritoneal dialysis that are living in a different county other than Jefferson county and has been on stable therapy for 2 months.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2015-04; Primary Completion 2020-11-17 (Actual); Study Completion 2020-11-17 (Actual)

PRIMARY OUTCOMES:
Change in Kidney Disease Quality Life Short Form 36 Survey when compared from the standard of care portion of the study to the telemedicine portion of the study | 36 months
  This outcome will determine the impact of telemedicine on quality of life as indicated two quality of life surveys.

SECONDARY OUTCOMES:
Composite endpoint of hospitalizations and peritonitis rates when comparing the time period on standard of care versus the time period of the telemedicine intervention. | 36 months
  Preliminary data will be obtained on rates of hospitalizations and peritonitis during participation in this study and compare from the standard of care portion of the study to the telemedicine portion of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Wallace, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States

REFERENCES:
- [Background] US Renal Data System: Bethesda, US Department of Public Health and Human Services, Public Health Service, National Institutes of Health, 2013
- [Background] Tonelli M, Hemmelgarn B, Culleton B, Klarenbach S, Gill JS, Wiebe N, Manns B; Alberta Kidney Disease Network. Mortality of Canadians treated by peritoneal dialysis in remote locations. Kidney Int. 2007 Oct;72(8):1023-8. doi: 10.1038/sj.ki.5002443. Epub 2007 Jul 18. PMID 17637709
- [Background] Nayak A, Karopadi A, Antony S, Sreepada S, Nayak KS. Use of a peritoneal dialysis remote monitoring system in India. Perit Dial Int. 2012 Mar-Apr;32(2):200-4. doi: 10.3747/pdi.2011.00124. No abstract available. PMID 22383718
- [Background] Afolalu B, Troidle L, Osayimwen O, Bhargava J, Kitsen J, Finkelstein FO. Technique failure and center size in a large cohort of peritoneal dialysis patients in a defined geographic area. Perit Dial Int. 2009 May-Jun;29(3):292-6. PMID 19458301
- [Background] Huisman RM, Nieuwenhuizen MG, Th de Charro F. Patient-related and centre-related factors influencing technique survival of peritoneal dialysis in The Netherlands. Nephrol Dial Transplant. 2002 Sep;17(9):1655-60. doi: 10.1093/ndt/17.9.1655. PMID 12198219
- [Background] Guo A, Mujais S. Patient and technique survival on peritoneal dialysis in the United States: evaluation in large incident cohorts. Kidney Int Suppl. 2003 Dec;(88):S3-12. doi: 10.1046/j.1523-1755.2003.08801.x. PMID 14870873
- [Background] Prakash S, Coffin R, Schold J, Lewis SA, Gunzler D, Stark S, Howard M, Rodgers D, Einstadter D, Sehgal AR. Travel distance and home dialysis rates in the United States. Perit Dial Int. 2014 Jan-Feb;34(1):24-32. doi: 10.3747/pdi.2012.00234. PMID 24525595
- [Background] Gallar P, Vigil A, Rodriguez I, Ortega O, Gutierrez M, Hurtado J, Oliet A, Ortiz M, Mon C, Herrero JC, Lentisco C. Two-year experience with telemedicine in the follow-up of patients in home peritoneal dialysis. J Telemed Telecare. 2007;13(6):288-92. doi: 10.1258/135763307781644906. PMID 17785025
- [Background] Nakamoto H, Hatta M, Tanaka A, Moriwaki K, Oohama K, Kagawa K, Wada K, Suzuki H. Telemedicine system for home automated peritoneal dialysis. Adv Perit Dial. 2000;16:191-4. PMID 11045291
- [Background] Lew SQ, Sikka N. Are patients prepared to use telemedicine in home peritoneal dialysis programs? Perit Dial Int. 2013 Nov-Dec;33(6):714-5. doi: 10.3747/pdi.2012.00203. No abstract available. PMID 24335134
- [Background] Fong E, Bargman JM, Chan CT. Cross-sectional comparison of quality of life and illness intrusiveness in patients who are treated with nocturnal home hemodialysis versus peritoneal dialysis. Clin J Am Soc Nephrol. 2007 Nov;2(6):1195-200. doi: 10.2215/CJN.02260507. Epub 2007 Oct 10. PMID 17928469
- [Background] Diamant MJ, Young A, Gallo K, Xi W, Suri RS, Garg AX, Moist LM. Hemodialysis in a satellite unit: clinical performance target attainment and health-related quality of life. Clin J Am Soc Nephrol. 2011 Jul;6(7):1692-9. doi: 10.2215/CJN.07650810. Epub 2011 May 12. PMID 21566106
- [Background] Samsa G, Edelman D, Rothman ML, Williams GR, Lipscomb J, Matchar D. Determining clinically important differences in health status measures: a general approach with illustration to the Health Utilities Index Mark II. Pharmacoeconomics. 1999 Feb;15(2):141-55. doi: 10.2165/00019053-199915020-00003. PMID 10351188